CLINICAL TRIAL: NCT00117572
Title: A Phase III Randomized Trial of Docetaxel Based Induction Chemotherapy in Patients With N2/N3 Locally Advanced Head and Neck Cancer
Brief Title: Docetaxel Based Chemotherapy Plus or Minus Induction Chemotherapy to Decrease Events in Head and Neck Cancer (DeCIDE)
Acronym: DeCIDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13362B
Record Dates: First submitted 2005-06-30; First posted 2005-07-07 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Cancer of the Pharynx; Cancer of the Larynx; Cancer of the Nasal Cavity; Paranasal Sinus Neoplasms; Cancer of the Oral Cavity
Keywords: Cancer of the Pharynx (Nasopharynx, Oropharynx, Hypopharynx); Cancer of the Nasal Cavity and Paranasal Sinuses
MeSH Terms: conditions — Pharyngeal Neoplasms; Laryngeal Neoplasms; Paranasal Sinus Neoplasms | interventions — Docetaxel; Cisplatin; Hydroxyurea; Fluorouracil; Drug Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Induction plus chemoradiotherapy (Active Comparator): Induction therapy: Two 21-day cycles of chemotherapy consisting of docetaxel (75 mg/m2, day 1), cisplatin (75 mg/m2, day 1), and 5-fluorouracil (750 mg/m2/day, days 1-5). Total duration of 6 weeks.
  Chemoradiotherapy: Five 14-day cycles of docetaxel (25 mg/m2, day 1), 5-fluorouracil (600 mg/m2/day, day 0-4), and hydroxyurea (500 mg PO q 12 hours x 6 days (11 doses)) with twice daily radiation (150 cGy given bid, days 1-5). Total duration of 10 weeks.
  Interventions: Drug: docetaxel; Drug: cisplatin; Drug: hydroxyurea; Drug: fluorouracil; Procedure: chemotherapy; Procedure: radiotherapy
- Chemoradiotherapy (Active Comparator): Chemoradiotherapy: Five 14-day cycles of docetaxel (25 mg/m2, day 1), 5-fluorouracil (600 mg/m2/day, day 0-4), and hydroxyurea (500 mg PO q 12 hours x 6 days (11 doses)) with twice daily radiation (150 cGy given bid, days 1-5). Total duration of 10 weeks.
  Interventions: Drug: docetaxel; Drug: hydroxyurea; Drug: fluorouracil; Procedure: chemotherapy; Procedure: radiotherapy

INTERVENTIONS:
Drug: docetaxel — 75 mg/m2 on day 1 (induction phase); 25 mg/m2 on day 1 (chemoradiotherapy phase)
Drug: cisplatin — 75 mg/m2 on day 1
  Arms: Induction plus chemoradiotherapy
Drug: hydroxyurea — Each cycle: 500 mg PO q 12 hours x 6 days (11 doses)
Drug: fluorouracil — 750 mg/m2/day on days 1-5 (induction phase); 600 mg/m2/day, day 0-4 (chemoradiotherapy phase)
Procedure: chemotherapy — See protocol for details
Procedure: radiotherapy — See protocol for details

SUMMARY:
The combined use of chemotherapeutic drugs with radiation has proven to be effective in improving overall survival and local control among patients with locally advanced head and neck cancer. Induction chemotherapy given before receiving local treatment has been shown to reduce the rate of distant failure. Many drugs have been found to prevent tumor cells from growing or dividing, although it has yet to be determined which agent, or specific combination of agents, is most effective in treating head and neck cancer. Docetaxel is a drug which has been reported to show promising activity in Phase II head and neck cancer studies. Therefore, the purpose of this trial is to compare the effectiveness of induction chemotherapy followed by chemoradiotherapy versus the same chemoradiotherapy alone in patients with locally advanced head and neck cancer.

DETAILED DESCRIPTION:
TRIAL DESIGN:

Phase III trial of induction therapy with docetaxel followed by chemoradiotherapy versus chemoradiotherapy alone in patients with nodal stage N2 or N3 head and neck cancer

OBJECTIVES:

Primary

* To determine the effect on overall survival when induction chemotherapy is administered prior to chemoradiotherapy in patients with N2 or N3 disease.

Secondary

* To determine the effect of induction chemotherapy when administered prior to chemoradiotherapy on distant failure-free survival, failure pattern, progression free survival and quality of life.

TREATMENT PLAN:

* After eligibility is confirmed, patients will be randomized to one of two treatment arms:

Arm A - Induction + chemoradiotherapy

Arm B - Chemoradiotherapy alone

* Induction therapy: Two 21-day cycles of chemotherapy consisting of docetaxel (day 1), cisplatin (day 1), and 5-fluorouracil (days 1-5). Total duration of 6 weeks.
* Chemoradiotherapy: Five 14-day cycles of docetaxel (day 1), 5-fluorouracil (day 0-4), and hydroxyurea (days 0-4) with twice daily radiation (days 1-5). Total duration of 10 weeks.
* All patients will undergo surgical evaluation after chemoradiation for possible neck dissection.
* Upon completion of treatment, patients will be monitored every three months during the first year, every six months during the second and third years, and annually thereafter, up to seven years.
* Patients will be followed for Quality of Life (QOL) during the course of treatment, as well as annually thereafter, up to five years.

PROJECTED ACCRUAL:

* An expected sample size of 400 patients will be enrolled for this study (200 per treatment arm).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Histologically or cytologically confirmed diagnosis of squamous cell or poorly differentiated carcinomas of the head and neck (excluding lip), or lymphoepithelioma
* No prior chemotherapy or radiotherapy
* Prior surgical therapy will consist only of incisional or excisional biopsy, and organ sparing procedures such as debulking of airway-compromising tumors or neck dissection in a patient with an existing primary tumor
* Karnofsky performance status of >= 70%
* Intact organ and bone marrow function
* Obtained informed consent

Exclusion Criteria:

* Demonstration of metastatic disease (i.e. M1 disease).
* Patients with a history of severe allergic reaction to docetaxel or other drugs formulated with polysorbate 80. History of allergic reactions attributed to compounds of similar chemical or biologic composition to cisplatin, 5-fluorouracil, or hydroxyurea
* Other coexisting malignancies or malignancies diagnosed within the previous 3 years with the exception of basal cell carcinoma, cervical cancer in situ, and other treated malignancies with no evidence of disease for at least 3 years.
* Prior surgical therapy other than incisional or excisional biopsy and organ-sparing procedures such as debulking of airway-compromising tumors or neck dissection in a patient with an unknown primary tumor. Any non-biopsy procedure must have taken place less than 3 months from initiating protocol treatment.
* Incomplete healing from previous surgery
* Pregnancy or breast feeding (men and women of child-bearing potential are eligible but must consent to using effective contraception during therapy and for at least 3 months after completing therapy)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (CHF), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with clinically significant pulmonary dysfunction, cardiomyopathy, or any history of clinically significant CHF are excluded. The exclusion of patients with active coronary artery disease will be at the discretion of the attending physician.
* Uncontrolled active infection unless curable with treatment of their cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2004-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everett Vokes, M.D., Principal Investigator — University of Chicago
Locations (26):
- United States (20):
  - USC University of Southern California Keck School of Medicine, Los Angeles, California
  - UM Sylvester Comprehensive Cancer Center, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Joliet Oncology Hematology Associates, Joliet, Illinois
  - Fort Wayne Medical Oncology/Hematology Inc., Fort Wayne, Indiana
  - AP&S Clinic, LLC, Terre Haute, Indiana
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Henry Ford Health System, Detroit, Michigan
  - Oncology Care Associates PLLC, Saint Joseph, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - UT Health Science Center at San Antonio, San Antonio, Texas
  - Oncology Alliance, Milwaukee, Wisconsin
- Croatia (2):
  - Clinic of Oncology, University Hospital Center Zagreb, Zagreb
  - University Hospital for Tumors Zagreb, Zagreb
- Clinique Armoricaine de Radiologie, Saint-Brieuc, France
- Russia (2):
  - NN Blokhin Russian Cancer Research Centre RAMS, Moscow
  - Republican Oncology Dispensary, Ufa
- Hospital Clínico San Carlos, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction Plus Chemoradiotherapy: Induction therapy: Two 21-day cycles of chemotherapy consisting of docetaxel (75 mg/m2, day 1), cisplatin (75 mg/m2, day 1), and 5-fluorouracil (750 mg/m2/day, days 1-5). Total duration of 6 weeks.
  Chemoradiotherapy: Five 14-day cycles of docetaxel (25 mg/m2, day 1), 5-fluorouracil (600 mg/m2/day, day 0-4), and hydroxyurea (500 mg PO q 12 hours x 6 days (11 doses)) with twice daily radiation (150 cGy given bid, days 1-5). Total duration of 10 weeks.
  docetaxel: 75 mg/m2 on day 1 (induction phase); 25 mg/m2 on day 1 (chemoradiotherapy phase)
  cisplatin: 75 mg/m2 on day 1
  hydroxyurea: Each cycle: 500 mg PO q 12 hours x 6 days (11 doses)
  fluorouracil: 750 mg/m2/day on days 1-5 (induction phase); 600 mg/m2/day, day 0-4 (chemoradiotherapy phase)
  chemotherapy: See protocol for details
  radiotherapy: See protocol for details
Period: Overall Study
Arm/Group | Induction Plus Chemoradiotherapy | Chemoradiotherapy
Started | 144 | 141
Completed | 138 | 135
Not Completed | 6 | 6
Not completed — Site withdrew before starting treatment | 2 | 3
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Induction Plus Chemoradiotherapy | Chemoradiotherapy | Total
Number analyzed (Participants) | 138 | 135 | 273
Age, Continuous [Mean (Full Range); unit: years] | 56.7 [31 to 75] | 56.9 [38 to 82] | 56.8 [31 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 17 | 42
  Male | 113 | 118 | 231
Region of Enrollment [Count of Participants; unit: Participants]
  France | 4 | 3 | 7
  United States | 120 | 123 | 243
  Spain | 1 | 0 | 1
  Croatia | 5 | 4 | 9
  Russia | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival: Time From Randomization to Death From Any Cause
Description: Survival rates over 6 years.
Time Frame: Up to 6 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Plus Chemoradiotherapy | Chemoradiotherapy
Number analyzed (Participants) | 138 | 135
percentage of participants | 74.9 [67.4 to 82.4] | 72.8 [65.1 to 80.6]
Statistical Analysis 1: Comparison: Induction Plus Chemoradiotherapy vs Chemoradiotherapy; Comparison of overall survival curves; Test type: Superiority or Other; p = 0.68, Log Rank; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.59 to 1.41] — Hazard ratio is (Induction+CRT)/CRT

2. Secondary Outcome: Distant Failure-free Survival (DFFS): Time From Randomization to Distant Recurrence or Death From Any Cause
Description: DFFS rates over 6 years. DFFS is time from randomization to distant recurrence or death from any cause
Time Frame: Up to 6 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Plus Chemoradiotherapy | Chemoradiotherapy
Number analyzed (Participants) | 138 | 135
percentage of participants | 69.3 [61.1 to 77.5] | 63.8 [55.4 to 72.2]
Statistical Analysis 1: Comparison: Induction Plus Chemoradiotherapy vs Chemoradiotherapy; Test type: Superiority or Other; p = 0.37, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.55 to 1.25] — Hazard ratio is (Induction+CRT)/CRT

3. Secondary Outcome: Recurrence Free Survival: Time From Randomization to Local/Regional/Distant Recurrence or Death From Any Cause
Description: Recurrence-free survival rates over 6 years. Recurrence-free survival is time from randomization to local, regional, or distant recurrence or death from any cause
Time Frame: Up to 6 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Plus Chemoradiotherapy | Chemoradiotherapy
Number analyzed (Participants) | 138 | 135
percentage of participants | 68.6 [60.6 to 76.7] | 58.6 [49.9 to 67.2]
Statistical Analysis 1: Comparison: Induction Plus Chemoradiotherapy vs Chemoradiotherapy; Test type: Superiority or Other; p = 0.16, Log Rank; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.51 to 1.12] — Hazard ratio is (Induction+CRT)/CRT

4. Secondary Outcome: Failure Pattern (Local/Regional Recurrence)
Description: Percentage of patients with local/regional recurrence
Time Frame: Up to 6 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Plus Chemoradiotherapy | Chemoradiotherapy
Number analyzed (Participants) | 138 | 135
percentage of participants | 10.1 [5.7 to 16.4] | 12.6 [7.5 to 19.4]
Statistical Analysis 1: Comparison: Induction Plus Chemoradiotherapy vs Chemoradiotherapy; Test type: Superiority or Other; p = 0.57, Fisher Exact

5. Secondary Outcome: Failure Pattern (Distant Recurrence)
Description: Percentage of patients with distant recurrence
Time Frame: Up to 6 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Plus Chemoradiotherapy | Chemoradiotherapy
Number analyzed (Participants) | 138 | 135
percentage of participants | 13.8 [8.5 to 20.7] | 21.5 [14.9 to 29.4]
Statistical Analysis 1: Comparison: Induction Plus Chemoradiotherapy vs Chemoradiotherapy; Test type: Superiority or Other; p = 0.11, Fisher Exact

6. Secondary Outcome: Quality of Life (FACT H&N)
Description: FACT Hand-and-neck subscale(b) (0-40 point scale with negative numbers indicating worsening of function)
Time Frame: Change from baseline to post-CRT (post-pre). This corresponds to week 16 in the induction arm and week 10 in the CRT alone arm.
Population: Survivors who completed the questionnaire. (Patients with missing data excluded.)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Induction Plus Chemoradiotherapy | Chemoradiotherapy
Number analyzed (Participants) | 77 | 85
units on a scale | -11.41 (1.11) | -12.34 (1.10)
Statistical Analysis 1: Comparison: Induction Plus Chemoradiotherapy vs Chemoradiotherapy; Test type: Superiority or Other; p = 0.55, t-test, 2 sided; Comparison of change scores between treatment groups

7. Secondary Outcome: Quality of Life (Normalcy of Diet)
Description: Performance Status Score (0-100 point scale with negative numbers indicating worsening of function)
Time Frame: as for outcome 6
Population: Survivors who completed the questionnaire. (Patients with missing data excluded.)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Induction Plus Chemoradiotherapy | Chemoradiotherapy
Number analyzed (Participants) | 75 | 86
units on a scale | -54.00 (3.95) | -41.51 (4.30)
Statistical Analysis 1: Comparison: Induction Plus Chemoradiotherapy vs Chemoradiotherapy; Test type: Superiority or Other; p = 0.034, t-test, 2 sided

8. Secondary Outcome: Quality of Life (Speech)
Description: Performance Status Score (0-100 point scale with negative numbers indicating worsening of function)
Time Frame: as for outcome 6
Population: Survivors who completed the questionnaire. (Patients with missing data excluded.)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Induction Plus Chemoradiotherapy | Chemoradiotherapy
Number analyzed (Participants) | 75 | 85
units on a scale | -10.67 (2.77) | -7.35 (2.21)
Statistical Analysis 1: Comparison: Induction Plus Chemoradiotherapy vs Chemoradiotherapy; Test type: Superiority or Other; p = 0.35, t-test, 2 sided

9. Secondary Outcome: Quality of Life (McMaster)
Description: McMaster RT Questionnaire (4-28 point scale with negative numbers indicating worsening of function)
Time Frame: as for outcome 6
Population: Survivors who completed the questionnaire. (Patients with missing data excluded.)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Induction Plus Chemoradiotherapy | Chemoradiotherapy
Number analyzed (Participants) | 76 | 84
units on a scale | -9.72 (0.90) | -9.79 (0.86)
Statistical Analysis 1: Comparison: Induction Plus Chemoradiotherapy vs Chemoradiotherapy; Test type: Superiority or Other; p = 0.96, t-test, 2 sided

10. Secondary Outcome: Quality of Life (FACT H&N)
Description: FACT Hand-and-neck subscale(b) (0-40 point scale with negative numbers indicating worsening of function)
Time Frame: Change from baseline to 1 year (1 year-pre)
Population: Survivors who completed the questionnaire. (Patients with missing data excluded.)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Induction Plus Chemoradiotherapy | Chemoradiotherapy
Number analyzed (Participants) | 43 | 40
units on a scale | -7.60 (1.14) | -7.34 (1.31)
Statistical Analysis 1: Comparison: Induction Plus Chemoradiotherapy vs Chemoradiotherapy; Test type: Superiority or Other; p = 0.88, t-test, 2 sided

11. Secondary Outcome: Quality of Life (Normalcy of Diet)
Description: Performance Status Score (0-100 point scale with negative numbers indicating worsening of function)
Time Frame: Change from baseline to 1 year (1 year-pre)
Population: Survivors who completed the questionnaire. (Patients with missing data excluded.)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Induction Plus Chemoradiotherapy | Chemoradiotherapy
Number analyzed (Participants) | 46 | 45
units on a scale | -10.22 (4.49) | -8.89 (4.09)
Statistical Analysis 1: Comparison: Induction Plus Chemoradiotherapy vs Chemoradiotherapy; Test type: Superiority or Other; p = 0.83, t-test, 2 sided

12. Secondary Outcome: Quality of Life (Speech)
Description: Performance Status Score (0-100 point scale with negative numbers indicating worsening of function)
Time Frame: Change from baseline to 1 year (1 year-pre)
Population: Survivors who completed the questionnaire. (Patients with missing data excluded.)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Induction Plus Chemoradiotherapy | Chemoradiotherapy
Number analyzed (Participants) | 44 | 44
units on a scale | -1.70 (1.70) | -3.41 (1.74)
Statistical Analysis 1: Comparison: Induction Plus Chemoradiotherapy vs Chemoradiotherapy; Test type: Superiority or Other; p = 0.49, t-test, 2 sided

13. Secondary Outcome: Quality of Life (McMaster)
Description: McMaster RT Questionnaire (4-28 point scale with negative numbers indicating worsening of function)
Time Frame: Change from baseline to 1 year (1 year-pre)
Population: Survivors who completed the questionnaire. (Patients with missing data excluded.)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Induction Plus Chemoradiotherapy | Chemoradiotherapy
Number analyzed (Participants) | 45 | 42
units on a scale | -3.29 (1.08) | -6.00 (1.15)
Statistical Analysis 1: Comparison: Induction Plus Chemoradiotherapy vs Chemoradiotherapy; Test type: Superiority or Other; p = 0.090, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 years
Arm/Group | Induction Plus Chemoradiotherapy | Chemoradiotherapy
All-Cause Mortality (participants affected / at risk) | 39/138 | 42/135
Serious Adverse Events (participants affected / at risk) | 65/138 | 38/135
Other Adverse Events (participants affected / at risk) | 132/138 | 129/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Plus Chemoradiotherapy (N=138) | Chemoradiotherapy (N=135)
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Agitation (Psychiatric disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 0
Ataxia (Nervous system disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bacteremia (Infections and infestations) | 5 | 1
Thromboembolic event (Vascular disorders) | 4 | 1
Hemorrhage (Blood and lymphatic system disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 — C-difficile
Cardiac stenosis (Cardiac disorders) | 1 | 0
Cellulitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Chills (General disorders) | 1 | 0
Confusion (Psychiatric disorders) | 2 | 1
Heart failure (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Death NOS (General disorders) | 3 | 1
Sepsis (Infections and infestations) | 3 | 2
Decreased PO intake (General disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 12 | 5
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 7 | 1
Dizziness (Nervous system disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 5 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Edema (General disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 1
Fatal bleeding (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 2
Fever (General disorders) | 14 | 9
Hallucinations (Psychiatric disorders) | 1 | 0
General status alteration (General disorders) | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Infection NOS (Infections and infestations) | 5 | 6
White blood cell decreased (Investigations) | 2 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 10 | 7
Nausea (Gastrointestinal disorders) | 5 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil count decreased (Investigations) | 8 | 0
Neutropenic fever (Investigations) | 6 | 0
Pain (General disorders) | 6 | 2
Peritoneal infection (Infections and infestations) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pulmonary MRI (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Reaction to vancomycin (Injury, poisoning and procedural complications) | 1 | 0
Pneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Positive staph aureus (Infections and infestations) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Syncope (Nervous system disorders) | 1 | 0
Throat pain (General disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Tracheostomy placement (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Vomiting (Gastrointestinal disorders) | 6 | 3
Weakness (General disorders) | 2 | 0
G-tube complications (Injury, poisoning and procedural complications) | 2 | 5
G-tube placement (Gastrointestinal disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Plus Chemoradiotherapy (N=138) | Chemoradiotherapy (N=135)
Fatigue (General disorders) | 118 | 94
Fever (General disorders) | 31 | 30
Alopecia (Skin and subcutaneous tissue disorders) | 63 | 34
Dermatitis radiation (Injury, poisoning and procedural complications) | 101 | 111
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 25 | 14 — Hand-foot skin reaction
Anorexia (Metabolism and nutrition disorders) | 85 | 75
Constipation (Gastrointestinal disorders) | 52 | 54
Dehydration (Metabolism and nutrition disorders) | 59 | 36
Diarrhea (Gastrointestinal disorders) | 62 | 31
Dysphagia (Gastrointestinal disorders) | 59 | 59
Mucositis oral (Gastrointestinal disorders) | 108 | 115
Nausea (Gastrointestinal disorders) | 91 | 72
Vomiting (Gastrointestinal disorders) | 59 | 40
Febrile neutropenia (Blood and lymphatic system disorders) | 22 | 2
Infection NOS (Infections and infestations) | 40 | 33
Edema limbs (General disorders) | 15 | 15
Neuropathy motor (Nervous system disorders) | 12 | 7
Neuropathy sensory (Nervous system disorders) | 20 | 8
Muscle pain (Musculoskeletal and connective tissue disorders) | 14 | 5
Headache (Nervous system disorders) | 12 | 10
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 48 | 44
Pain (General disorders) | 61 | 64
Neutrophil count decreased (Investigations) | 83 | 36
Hemoglobin (Investigations) | 127 | 123
Platelet count decreased (Investigations) | 56 | 34
Hyperglycemia (Metabolism and nutrition disorders) | 121 | 113
Hypoglycemia (Investigations) | 17 | 13
White blood cell decreased (Investigations) | 117 | 89
Aspartate aminotransferase increased (Investigations) | 43 | 45
Alanine aminotransferase increased (Investigations) | 55 | 59
Alkaline phosphatase increased (Investigations) | 60 | 27
Blood bilirubin increased (Investigations) | 19 | 12
Creatinine increased (Investigations) | 37 | 16
Anxiety (Psychiatric disorders) | 12 | 12
Candidiasis (Infections and infestations) | 13 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 14
Depression (Psychiatric disorders) | 15 | 9
Dizziness (Nervous system disorders) | 15 | 5
Dry mouth (Gastrointestinal disorders) | 24 | 26
Dysgeusia (Nervous system disorders) | 13 | 13
Dyspepsia (Gastrointestinal disorders) | 11 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 16 | 12
Hypocalcemia (Metabolism and nutrition disorders) | 22 | 15
Hypokalemia (Metabolism and nutrition disorders) | 29 | 14
Hypomagnesemia (Metabolism and nutrition disorders) | 23 | 8
Hyponatremia (Metabolism and nutrition disorders) | 26 | 14
Hypotension (Vascular disorders) | 8 | 3
Insomnia (Psychiatric disorders) | 12 | 11
Lymphocyte count decreased (Investigations) | 6 | 9
Odynophagia (Gastrointestinal disorders) | 7 | 9
Oral candidiasis (Infections and infestations) | 9 | 6
Oral pain (Gastrointestinal disorders) | 11 | 9
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Stomatitis (Gastrointestinal disorders) | 13 | 6
Weight loss (Investigations) | 32 | 27
Late RT - Esophagus (Gastrointestinal disorders) | 13 | 11 — Late event--after completion of therapy.
Late RT - Larynx (Gastrointestinal disorders) | 7 | 5 — Late event--after completion of therapy.
Late RT - Mucous membrane (Gastrointestinal disorders) | 19 | 21 — Late event--after completion of therapy.
Late RT - Salivary glands (Gastrointestinal disorders) | 24 | 25 — Late event--after completion of therapy.
Late RT - Skin (Skin and subcutaneous tissue disorders) | 15 | 18
Late RT - Anoxrexia (Metabolism and nutrition disorders) | 10 | 14 — Late event--after completion of therapy.
Late - Constipation (Gastrointestinal disorders) | 7 | 5 — Late event--after completion of therapy.
Late - Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 3 — Late event--after completion of therapy.
Late - Dry mouth (Gastrointestinal disorders) | 47 | 46 — Late event--after completion of therapy.
Late - Dysphagia (Gastrointestinal disorders) | 24 | 33 — Late event--after completion of therapy.
Late - Fatigue (General disorders) | 19 | 25 — Late event--after completion of therapy.
Late - Mucosal inflammation (Gastrointestinal disorders) | 11 | 6 — Late event--after completion of therapy.
Late - Oral pain (Gastrointestinal disorders) | 9 | 1 — Late event--after completion of therapy.
Late - Pain (General disorders) | 10 | 14 — Late event--after completion of therapy.
Late - Weight loss (Investigations) | 7 | 5 — Late event--after completion of therapy.
Late - Dysgeusia (Nervous system disorders) | 9 | 11 — Late event--after completion of therapy.
Trismus (Musculoskeletal and connective tissue disorders) | 3 | 8 — Late event--after completion of therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes